CLINICAL TRIAL: NCT07300098
Title: Epidemiological Evaluation of Knee Injuries in Children Admitted to Assiut University Hospitals From 2022 to 2025.
Status: Active, not recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mohamed Mahmoud Ebrahim Abd Allah, MMEAAllah, Assiut University
Other Study IDs: evaluation of knee injuries
Record Dates: First submitted 2025-12-10; First posted 2025-12-23 (Actual); Last update posted 2025-12-23 (Actual); Status verified 2025-12

CONDITIONS: Knee Injuries
Keywords: knee injuries
MeSH Terms: conditions — Knee Injuries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 10 Weeks
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
To categorize and analyze the incidence of the knee injuries in children admitted in Assiut University from 2022 to 2025 and to establish a data base about children less than 18 years who have knee injuries for further studies.

DETAILED DESCRIPTION:
Knee injuries are common in children and constitute about 5 %of the injuries presenting to emergency department in 1 to 18 y age group . The presence of physis or growth plate, which is weaker compared to the adjacent ligaments make injury patterns in children different from those in adults, as the same amount of force would produce a physeal fracture or avulsion injury in children but a ligament injury in an adult.

Kraus et al. divided patients according to age to infants (younger than 1 year); pre-school aged children (1-6 years); prepubertal school-aged children (7-10 years); early adolescent patients (11-14 years); late adolescent patients (15-18 years) and a five diagnosis-related groups : extraarticular soft tissue injuries, intraarticular soft tissue injuries, patella disorders, fractures, and overload injuries. They found extraarticular soft tissue injuries were most common and fractures were rare.

Skak et al found that children with ligament injuries and physeal fractures had a median age of 12 years. No lesions of the cruciate ligaments without bony avulsion were diagnosed. the most frequent cause of injuries was falls.

The most frequent traumatic injuries reported involve the cruciate and collateral ligaments (medial collateral ligament [MCL], posterior cruciate ligament [PCL], anterior cruciate ligament [ACL], and lateral collateral ligament [LCL]), menisci, and patella. Overall, females are reported to have a higher risk of sustaining a knee injury than males. Ligament injuries ,specifically ACL injuries, are among the most devastating knee injuries for young patients. Female patients have two to eight times greater risk of sustaining an ACL injury as compared with male patients. After ACL injury, there is a significant risk of developing osteoarthritis regardless of the treatment intervention, such as ACL on surgery.

The rationale of the research is to establish a data base about children less than 18 years who have knee injuries for further studies.

research and injury pattern analysis. All imaging studies stored in PACS and the operative notes and clinical data documented will be verified to enhance data validity and completeness.

The data collection process will not be limited to basic demographic and diagnostic variables. A comprehensive data abstraction form will be developed to ensure standardized retrieval of relevant clinical presentation, radiological, and final management of the patients. The extracted data will include mechanism and date of trauma, anatomical injury characteristics, associated injuries, type of management (conservative or operative), intra-operative details when applicable, radiological findings.

2.4.5 -Research outcome measures:

1. Primary (main):

   The epidemiology (incidence and patterns) of knee injuries among children (<18 years) admitted to Assiut University Hospitals between 2022 and 2025 to establish a data base about children less than 18 years who have knee injuries for further studies .and all extracted data and radiological images will be securely entered into a password-protected, anonymized electronic database (such as Red cap) to ensure confidentiality, facilitate statistical analysis, and allow future reference by the research team in compliance with institutional ethical standards.
2. Secondary (subsidiary): none

ELIGIBILITY:
Inclusion Criteria:

* Children admitted with knee injuries (open or closed) in Assiut University.

Exclusion Criteria:

* No

Ages: 1 Year to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Children admitted with knee injuries (open or closed) in Assiut University.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2025-12-10 (Actual); Primary Completion 2026-01-01 (Estimated); Study Completion 2026-01-01 (Estimated)

PRIMARY OUTCOMES:
establish a data base about children less than 18 years who have knee injuries for further studies | between 2022 and 2025
  The epidemiology (incidence and patterns) of knee injuries among children (<18 years) admitted to Assiut University Hospitals between 2022 and 2025 to establish a data base about children less than 18 years who have knee injuries for further studies .and all extracted data and radiological images will be securely entered into a password-protected, anonymized electronic database (such as Red cap) to ensure confidentiality, facilitate statistical analysis, and allow future reference by the research team in compliance with institutional ethical standards.

CONTACTS AND LOCATIONS:
Overall Officials: Nariman Abol Oyoun, associated prof, Study Chair — Assiut University; Hatem Galal El-Din Zaki, prof, Study Chair — Assiut University
Locations (1):
- Assuit University, Asyut, Ass, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] O'Kane JW, Neradilek M, Polissar N, Sabado L, Tencer A, Schiff MA. Risk Factors for Lower Extremity Overuse Injuries in Female Youth Soccer Players. Orthop J Sports Med. 2017 Oct 23;5(10):2325967117733963. doi: 10.1177/2325967117733963. eCollection 2017 Oct. PMID 29114563
- [Result] Arnold A, Thigpen CA, Beattie PF, Kissenberth MJ, Shanley E. Overuse Physeal Injuries in Youth Athletes. Sports Health. 2017 Mar/Apr;9(2):139-147. doi: 10.1177/1941738117690847. Epub 2017 Feb 6. PMID 28165873
- [Result] Swenson DM, Collins CL, Best TM, Flanigan DC, Fields SK, Comstock RD. Epidemiology of knee injuries among U.S. high school athletes, 2005/2006-2010/2011. Med Sci Sports Exerc. 2013 Mar;45(3):462-9. doi: 10.1249/MSS.0b013e318277acca. PMID 23059869
- [Result] Butler LS, Janosky JJ, Sugimoto D. Pediatric and Adolescent Knee Injuries: Risk Factors and Preventive Strategies. Clin Sports Med. 2022 Oct;41(4):799-820. doi: 10.1016/j.csm.2022.05.011. PMID 36210172
- [Result] Skak SV, Jensen TT, Poulsen TD, Sturup J. Epidemiology of knee injuries in children. Acta Orthop Scand. 1987 Feb;58(1):78-81. doi: 10.3109/17453678709146348. PMID 3577744
- [Result] Kraus T, Svehlik M, Singer G, Schalamon J, Zwick E, Linhart W. The epidemiology of knee injuries in children and adolescents. Arch Orthop Trauma Surg. 2012 Jun;132(6):773-9. doi: 10.1007/s00402-012-1480-0. Epub 2012 Feb 23. PMID 22358221
- [Result] Parikh SN, Shrivastava RK. Evaluation of Children with Injuries Around the Knee. Indian J Pediatr. 2016 Aug;83(8):844-51. doi: 10.1007/s12098-015-1993-y. Epub 2016 Feb 29. PMID 26924653